CLINICAL TRIAL: NCT05378542
Title: Evaluation of the Efficiency of Nursing Care Given Through the Mobil Health Application Developed for Cervical Cancer.
Brief Title: Mobile Health Application Developed for Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Associate professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 006scltnmn
Record Dates: First submitted 2022-04-21; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: MOBİLE HEALTH, CERVİCAL CANCER, AWARENESS
MeSH Terms: conditions — Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: The research is a single center, parallel group, stratified block randomized controlled experimental study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Stratified block randomization will be used to avoid selection bias. In this study on application bias, researcher and participant blinding will not be done. Because the researcher will make the application himself and placebo cannot be used in the intervention.
  Data collection forms to prevent detection bias will be applied online through Google Forms® independently of the researcher.
  The data obtained from the research aimed at preventing reporting bias will be coded as A and B by an independent researcher and transferred to the SPSS program. Analysis of the data will also be done by an independent statistician.
  In order to prevent attrition bias, Intention to Treat Test will be used in the sample group in case of missing/subtracting or not completing the post-tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. group (Active Comparator): participants will receive information about cervical cancer with the developed mobile application.
  Interventions: Behavioral: Mobile application usage
- 2. group (No Intervention): No Intervention: control group (non-education) Routıne care

INTERVENTIONS:
Behavioral: Mobile application usage — The implementation of the research was carried out in two stages. In the first stage, a mobile application was created, in the second stage, training and counseling was given to the experimental group with the mobile application, and no attempt was made to the control group.
  Arms: 1. group

SUMMARY:
The main purpose of this research is to evaluate the effect of the nursing care that participants receive with the mobile health application for cervical cancer on raising awareness about cervical cancer. The study conducted through the mobile health application developed to raise awareness about cervical cancer; It is thought that it is important in terms of raising awareness of participants, easing the work-time burden of health personnel in this period, and reducing the cost of health care through early diagnosis and treatment, and will set an example for future studies. Positive outputs from the mobile application will allow the application to be used on national and international platforms.

DETAILED DESCRIPTION:
In the face-to-face health care system, especially due to the pandemic period, the problem of personnel need to provide health care can be solved with mobile health applications; thus, mobile health applications can indirectly help workforce problems. Mobile applications allow the provision of high quality, useful services with less energy and cost to large audiences. In addition, mobile health applications allow patients to be followed remotely, allowing patients to access health services wherever, whenever and as often as they want. It is stated that well-structured mobile applications have a positive impact on the health sector. In this context, it is seen that the use of mobile applications in primary, secondary and tertiary healthcare services is becoming increasingly common all over the world.

In researches planned study, it is aimed to develop a mobile application in Turkish in order to raise awareness about cervical cancer and to evaluate its effectiveness. In the content of the mobile application to be developed, information about cervical cancer such as information about cervical cancer, symptoms, findings, diagnosis, screening, treatment, practical explanations with video, frequently asked questions about the subject; It is planned to have interim notifications, reminders, pay attention warning messages. There are a limited number of practices related to cervical cancer awareness in the world. In Turkey, there is no e-health mobile application for cervical cancer awareness. Unlike the applications in the world; In the application, which is aimed to be developed in this study, there is an area where the participants can ask questions to the researcher from the "Request Support" section and there is a field. The information provided by mobile health applications was found to be educational, appropriate, original and on-site, and it was found useful to be reliable. Studies have shown that mobile health applications contribute to positive health outcomes.

The study conducted through the mobile health application developed to raise awareness about cervical cancer; It is thought that it is important in terms of raising the awareness of participants, easing the work-time burden of health personnel in this period, and reducing the cost of health care through early diagnosis and treatment, and will set an example for future studies. Positive outputs from the mobile application will allow the application to be used on national and international platforms.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 and over
* Able to understand and speak Turkish
* ability to read and write
* Owning a smartphone

Exclusion Criteria:

* Having a communication barrier (seeing, understanding...)
* Having been diagnosed with cervical cancer in himself or his first degree relatives
* Not wanting to leave work
* the lost of life,
* Not participating in the final tests,
* Failure to complete parts of the mobile application within the specified time,

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Mobile Health Application questionnaire: "There is "NO" difference in the mean scores of Cervical Cancer and Pap Smear Test Health Belief Model Scale between women who received | 2 months
  In the nursing care given with the mobile health application for cervical cancer, in the experimental and control groups
Mobile Health Application questionnaire: "There is "YES' difference in the mean scores of Cervical Cancer and Pap Smear Test Health Belief Model Scale between women who received | 2 months
  the nursing care given with the mobile health application for cervical cancer, in the experimental and control groups

CONTACTS AND LOCATIONS:
Overall Officials: seçil güneysu tunaman, Principal Investigator — bursa provincial health directorate
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No